CLINICAL TRIAL: NCT02709161
Title: Effects of Amygdala Neurofeedback on Depressive Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The grant funding ran out
Sponsor: Kymberly Young (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Kymberly Young, Assistant Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19110101; R00MH101235 (NIH)
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder
Keywords: neurofeedback; major depressive disorder; amygdala
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- real-time fMRI neurofeedback: Amygdala (Experimental): Amygdala neurofeedback - attempt to upregulate the left amygdala during positive autobiographical memory recall via real time fMRI neurofeedback from the amygdala. Two sessions will be performed one week apart.
  Interventions: Device: real-time fMRI neurofeedback: Amygdala
- real-time fMRI neurofeedback: HIPS (Active Comparator): HIPS neurofeedback - attempt to upregulate the left horizontal segment of the intraparietal sulcus (HIPS), a region not involved in emotional processing, during positive autobiographical memory recall via real time fMRI neurofeedback from the HIPS. Two sessions will be performed one week apart.
  Interventions: Device: real-time fMRI neurofeedback: HIPS

INTERVENTIONS:
Device: real-time fMRI neurofeedback: Amygdala — Participants are shown activity from their left amygdala in real time and are instructed to increase the level of activity in that region by thinking of positive autobiographical memories
  Arms: real-time fMRI neurofeedback: Amygdala
Device: real-time fMRI neurofeedback: HIPS — Participants are shown activity from their left horizontal segment of the intraparietal sulcus in real time and are instructed to increase the level of activity in that region by thinking of positive autobiographical memories
  Arms: real-time fMRI neurofeedback: HIPS

SUMMARY:
The purpose of this study is to determine the clinical efficacy of augmenting cognitive-behavioral therapy with real-time functional magnetic resonance imaging neurofeedback (rtfMRI-nf) training to increase the amygdala's response to positive autobiographical memories.

DETAILED DESCRIPTION:
Previous research has shown that real-time fMRI neurofeedback (rtfMRI-nf) training aimed at increasing the amygdala's response to positive autobiographical memory recall holds therapeutic potential for treating patients with major depressive disorder (MDD), as clinically significant decreases in clinician administered and self-report measures of depression severity were observed following two rtfMRI amygdala neurofeedback sessions. Furthermore, rtfMRI amygdala neurofeedback changed emotional processing towards a positive bias. As this rtfMRI-nf procedure utilizes principles of cognitive-behavioral therapy (CBT), including restructuring thoughts and emotional processing towards the positive, the current study seeks to examine the effects of augmenting CBT with amygdala rtfMRI-nf. Specifically, the investigators plan to test the hypothesis that pretreatment with two amygdala rtfMRI-nf sessions prior to the the start of CBT will result in a higher percentage of patients who exhibit 'sudden gains' (a between session drop of at least 25% on the Beck Depression Inventory associated with better treatment response) compared to those who receive rtfMRI-nf from a parietal control region putatively not involved in emotional processing. Over the course of three years, 60 participants diagnosed with MDD and planning to start CBT will be recruited through the clinical services of the Western Psychiatric Institute and Clinic (WPIC) and through licensed CBT therapists in the Pittsburgh metropolitan area. Participants will undergo two rtfMRI-nf sessions within the two weeks prior to starting therapy. Half of the participants will receive amygdala neurofeedback and half will receive control neurofeedback. At weeks 1-3 and 9 & 10 following the start of therapy, the participant will complete the BDI-II and the NIH Patient Reported Outcomes Measurement Information System (PROMIS) Depression measure. The number of patients who meet criteria for sudden gains and the average session at which this occurred will be compared between CBT + amygdala rtfMRI-nf and CBT + control rtfMRI-nf groups. Success will suggest a new method for improving outcomes to CBT in depressed patients.

ELIGIBILITY:
Inclusion Criteria:

* right-handed adults
* ages 18 - 55
* primary diagnosis of MDD for recurrent MDD who are currently depressed
* able to give written informed consent prior to participation
* unmedicated OR are stable on an unsuccessful antidepressant regime (at least 4 weeks to ensure symptoms are stable). Effective medications will not be discontinued for the purposes of the study.

Exclusion Criteria:

* clinically significant or unstable cardiovascular, pulmonary, endocrine, neurological, gastrointestinal illness or unstable medical disorder
* alcohol and/or substance dependence (other than nicotine) within 12 months prior to screening
* history of traumatic brain injury
* unable to complete MRI scan due to claustrophobia or general MRI exclusions (e.g., shrapnel inside body)
* currently pregnant or breast feeding
* unable to complete questionnaires written in English
* current (within 3 weeks of testing) use of any antipsychotics, anticonvulsants, stimulants, benzodiazepines, beta-blockers, or other medications (except antidepressants) likely to influence cerebral blood flow. Effective medications will not be discontinued for the purposes of the study. I
* diagnosis of psychotic or organic mental disorder, bipolar I or II disorder.
* eye problems or difficulties in corrected vision.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Compere L, Siegle GJ, Lazzaro S, Strege M, Canovali G, Barb S, Huppert T, Young K. Real-time functional magnetic resonance imaging neurofeedback training of amygdala upregulation increases affective flexibility in depression. J Psychiatry Neurosci. 2023 Jun 20;48(3):E232-E239. doi: 10.1503/jpn.220208. Print 2023 May-Jun. PMID 37339817

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real-time fMRI Neurofeedback: Amygdala | Real-time fMRI Neurofeedback: HIPS
Started | 19 | 17
Completed | 18 | 17
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real-time fMRI Neurofeedback: Amygdala | Real-time fMRI Neurofeedback: HIPS | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (12) | 31 (9) | 32 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 18 | 15 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36
Beck Depression Inventory Baseline [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory is a self-report questionnaire consisting of 21 questions assessing depressive symptoms. Scores can range from 0-63 with higher scores indicating more severe depression.
  units on a scale | 27.2 (10.7) | 26.6 (13.4) | 26.8 (11.8)
PROMIS Baseline [Mean (Standard Deviation); unit: t-score] — The PROMIS depression measure is a self-report measure of depressive symptoms consisting of 8 questions. Scores can range from 0-40 with higher scores indicating greater severity of depression. The raw scores are converted to T scores with a mean of 50 and standard deviation of 10. Scores under 55 indicate no depression and scores above 70 indicating severe depression.
  t-score | 68 (8) | 66 (9) | 67 (9)

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory (BDI-II)
Description: The Beck Depression Inventory is a self-report questionnaire consisting of 21 questions assessing depressive symptoms. Scores can range from 0-63 with higher scores indicating more severe depression.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real-time fMRI Neurofeedback: Amygdala | Real-time fMRI Neurofeedback: HIPS
Number analyzed (Participants) | 18 | 15
units on a scale | 16.1 (9.66) | 24.3 (12.3)
Statistical Analysis 1: Comparison: Real-time fMRI Neurofeedback: Amygdala vs Real-time fMRI Neurofeedback: HIPS; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = 8.2

2. Secondary Outcome: PROMIS Item Bank v1.0 - Depression
Description: The PROMIS depression measure is a self-report measure of depressive symptoms consisting of 8 questions. Scores can range from 0-40 with higher scores indicating greater severity of depression. The raw scores are converted to T scores with scores with a mean of 50 and a standard deviation of 10. Scores under 55 indicate no depression and scores above 70 indicate severe depression.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Real-time fMRI Neurofeedback: Amygdala | Real-time fMRI Neurofeedback: HIPS
Number analyzed (Participants) | 18 | 15
t-score | 53 (11) | 61 (12)
Statistical Analysis 1: Comparison: Real-time fMRI Neurofeedback: Amygdala vs Real-time fMRI Neurofeedback: HIPS; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = 8.2

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Real-time fMRI Neurofeedback: Amygdala | Real-time fMRI Neurofeedback: HIPS
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT02709161/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT02709161/ICF_001.pdf